CLINICAL TRIAL: NCT06740630
Title: A Phase 3a, Observer-blind, Randomized, Controlled Study to Demonstrate Lot-to-lot Consistency and Evaluate the Immunogenicity and Safety of an Investigational Varicella Vaccine Compared With Varivax, Administered as a First Dose to Healthy Children 12 to 15 Months of Age
Brief Title: A Study on the Immune Response and Safety of an Investigational Chickenpox Vaccine When Given to Healthy Children 12 to 15 Months of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 213998; 2024-515869-33-00 (Other: EU CT Number)
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chickenpox
Keywords: Chicken pox; VNS; Varicella; Varivax; Healthy Children
MeSH Terms: conditions — Chickenpox | interventions — Measles-Mumps-Rubella Vaccine; Hepatitis A Vaccines; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Observer-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- VNS_Lot 1 Group (Experimental): Participants receive 1 dose of the investigational VNS vaccine of Lot 1, 1 dose of measles, mumps, and rubella (MMR) vaccine, 1 dose of hepatitis A vaccine (HAV), and 1 dose of PCV (either PCV 13 or Vaxneuvance or PCV 20) on Day 1.
  Interventions: Biological: Investigational varicella vaccine_Lot 1; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance
- VNS_Lot 2 Group (Experimental): Participants receive 1 dose of the investigational VNS vaccine of Lot 2, 1 dose of MMR vaccine, 1 dose of HAV vaccine, and 1 dose of PCV (either PCV 13 or Vaxneuvance or PCV 20) on Day 1.
  Interventions: Biological: Investigational varicella vaccine_Lot 2; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance
- VNS_Lot 3 Group (Experimental): Participants receive 1 dose of the investigational VNS vaccine of Lot 3, 1 dose of MMR vaccine, 1 dose of HAV vaccine, and 1 dose of PCV (either PCV 13 or Vaxneuvance or PCV 20) on Day 1.
  Interventions: Biological: Investigational varicella vaccine_Lot 3; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance
- VV_Lot 1 Group (Active Comparator): Participants receive 1 dose of a marketed varicella vaccine (VV) of Lot 1, 1 dose of MMR vaccine, 1 dose of HAV vaccine, and 1 dose of PCV (either PCV 13 or Vaxneuvance or PCV 20) on Day 1.
  Interventions: Biological: Marketed varicella vaccine_Lot 1; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance
- VV_Lot 2 Group (Active Comparator): Participants receive 1 dose of a marketed VV of Lot 2, 1 dose of MMR vaccine, 1 dose of HAV vaccine, and 1 dose of PCV (either PCV 13 or Vaxneuvance or PCV 20) on Day 1.
  Interventions: Biological: Marketed varicella vaccine_Lot 2; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance

INTERVENTIONS:
Biological: Investigational varicella vaccine_Lot 1 — Investigational varicella vaccine of Lot 1 administered subcutaneously.
  Arms: VNS_Lot 1 Group
Biological: Investigational varicella vaccine_Lot 2 — Investigational varicella vaccine of Lot 2 administered subcutaneously.
  Arms: VNS_Lot 2 Group
Biological: Investigational varicella vaccine_Lot 3 — Investigational varicella vaccine of Lot 3 administered subcutaneously.
  Arms: VNS_Lot 3 Group
Biological: Marketed varicella vaccine_Lot 1 — Marketed varicella vaccine of Lot 1 administered subcutaneously.
  Arms: VV_Lot 1 Group
Biological: Marketed varicella vaccine_Lot 2 — Marketed varicella vaccine of Lot 2 administered subcutaneously.
  Arms: VV_Lot 2 Group
Biological: MMR vaccine — MMR vaccine co-administered subcutaneously or intramuscularly.
Biological: Hepatitis A vaccine — Hepatitis A vaccine co-administered intramuscularly.
Biological: PCV (pneumococcal conjugate vaccine) 13 — The 13-valent pneumococcal conjugate vaccine co-administered intramuscularly. In some countries PCV will only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.
Biological: PCV 20 — The 20-valent pneumococcal conjugate vaccine co-administered intramuscularly. In some countries PCV will only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.
Biological: Vaxneuvance — The Vaxneuvance (15-valent pneumococcal conjugate vaccine) co-administered intramuscularly. In some countries PCV will only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.

SUMMARY:
The purpose of this study is to assess the consistency of immune response to three different lots of GSK's investigational varicella vaccine (VNS Vaccine), and to compare the safety and immune response of VNS vaccine to an already approved varicella vaccine (VV) known as Varivax. The study will be conducted in healthy children aged 12 to 15 months, who have neither contracted varicella nor received a varicella vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent(s) Legally acceptable representatives /(LAR[s]), who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiaries, return for follow-up visits).
* Written or witnessed/thumb printed informed consent obtained from the participant's parent(s)/LAR(s) prior to performance of any study-specific procedure.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female between, and including, 12 to 15 months of age (i.e., from the day of 1-year birthday until the day before 16 months of age) at the time of the administration of study interventions.
* Only for children in countries where PCV is recommended at 12 to 15 months of age as per national immunization schedule and provided as part of the study interventions:

  * Participant who previously received the primary series of PCV in the first year of life with last dose at least 60 days prior to study entry.

Exclusion Criteria:

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hypersensitivity to latex.
* Major congenital defects, as assessed by the investigator.
* Recurrent history of uncontrolled neurological disorders or seizures.
* History of varicella disease.
* Active untreated tuberculosis.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study interventions during the period beginning 30 days before the dose of study interventions administration (Day -29 to Day 1), or their planned use during the study period.
* Planned administration of a vaccine in the period starting 30 days before the dose and ending 43 days after the dose of study interventions administration* (Visit 2) with the exception of inactivated influenza vaccine which may be given at any time during the study and administered at a different location than the study interventions.

Any other age-appropriate vaccine may be given starting at Visit 2 and anytime thereafter.

*If emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is organized by public health authorities outside the routine immunization program, the time period described above can be reduced provided it is used according to the local governmental recommendations and sponsor is notified

* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune modifying treatments at any time up to the end of the study.

  * Up to 90 days prior to the study intervention administration:
  * For corticosteroids, this will mean prednisone equivalent >=0.5 mg/kg/day with maximum of 20 mg/day for pediatric participants. Inhaled and topical steroids are allowed.
  * Administration of immunoglobulins and/or any blood products or plasma derivatives.
  * Up to 180 days prior to study interventions administration: long acting immune-modifying drugs including among others immunotherapy (e.g., tumor necrosis factor-inhibitors), monoclonal antibodies (except the ones not interfering with the immune response to the study vaccines, e.g., nirsevimab), antitumoral medication.
* Previous vaccination against measles, mumps, and rubella.
* Previous vaccination against hepatitis A virus.
* Previous vaccination against varicella virus.
* Only for children in countries where PCV is recommended at 12 to 15 months of age as per national immunization schedule and provided as part of the study interventions, participant who previously received a booster dose of any PCV.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).
* Child in care.
* Any study personnel's immediate dependents, family, or household members.
* Participants with the following high-risk individuals in their household:

  * Immunocompromised individuals.
  * Pregnant women without documented history of varicella.
  * Newborn infants of mothers without documented history of varicella.
  * Newborn infants born less than (<) 28 weeks of gestation.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1840 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-05-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with seroresponse to Varicella Zoster Virus (VZV) anti-glycoprotein E (gE) Immunoglobulin (IgG) for the 3 lots of VNS vaccine groups | At Day 43
  Seroresponse is defined as post-vaccination (Day 43) anti-VZV gE IgG antibody concentration greater than or equal to (>=) 300 milli-international units per milliliter (mIU/mL) among participants who were seronegative [(antibody concentration less than (<) LLOQ (Lower limit of quantification)] before vaccination. A seronegative participant is a participant whose antibody concentration is below the LLOQ of the assay. A seropositive participant is a participant whose antibody concentration is greater than or equal to the LLOQ of the assay.
Geometric Mean Concentration (GMC) of anti-VZV gE IgG for the 3 lots of VNS vaccine groups | At Day 43
  Concentrations of anti-VZV gE IgG presented as GMCs and expressed in mIU/mL for each group.
Percentage of participants with seroresponse to anti-VZV gE IgG for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups | At Day 43
  Seroresponse is defined as post-vaccination (Day 43) anti-VZV gE IgG concentration >= 300 mIU/mL among participants who were seronegative (antibody concentration < LLOQ) before vaccination. A seronegative participant is a participant whose antibody concentration is below the LLOQ of the assay. A seropositive participant is a participant whose antibody concentration is greater than or equal to the LLOQ of the assay.
GMCs of anti-VZV gE IgG for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups | At Day 43
  Concentrations of anti-VZV gE IgG are presented as GMCs and expressed in mIU/mL for each group.

SECONDARY OUTCOMES:
Anti-measles antibodies GMCs for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups | At Day 43
Anti-mumps antibodies GMCs for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups | At Day 43
Anti-rubella antibodies GMCs for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups | At Day 43
Percentage of participants with seroresponse to anti-measles for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups | At Day 43
  Seroresponse is defined as post-vaccination (Day 43) anti-measles antibody concentration >= cut-off value among participants who were seronegative (antibody concentration < cut-off value) before vaccination.
  The assay cut-off values for anti-measles will be defined by the laboratory before the analysis.
Percentage of participants with seroresponse to anti-mumps for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups | At Day 43
  Seroresponse is defined as post-vaccination (Day 43) anti-mumps antibody concentration >= cut-off value among participants who were seronegative (antibody concentration < cut-off value) before vaccination.
  The assay cut-off values for anti-mumps will be defined by the laboratory before the analysis.
Percentage of participants with seroresponse to anti-rubella for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups | At Day 43
  Seroresponse is defined as post-vaccination (Day 43) anti-rubella antibody concentration >= cut-off value among participants who were seronegative (antibody concentration < cut-off value) before vaccination.
  The assay cut-off values for anti-rubella will be defined by the laboratory before the analysis.
Anti-Hepatitis A antibodies GMCs for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups in Hepatitis A virus (HAV) subset | At Day 43
Percentage of participants with seroresponse to anti-HAV for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups in HAV subset | At Day 43
  Seroresponse is defined as post-vaccination (Day 43) anti-HAV antibody concentration >= cut-off value among participants who were seronegative (antibody concentration < cut-off value) before vaccination.
  The assay cut-off values for anti-HAV antibodies will be defined by the laboratory before the analysis.
Anti-S. pneumoniae serotype specific Polysaccharide IgG antibody concentrations for the 3 pooled lots of VNS vaccine groups compared with the 2 pooled lots of VV groups in PCV subset | At Day 43
  S. pneumoniae polysaccharides to be tested: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F.
Percentage of participants in the VNS vaccine pooled group with anti-VZV gE antibody concentrations above the adaptive seroresponse threshold | At Day 43
  The adaptive seroresponse threshold is the anti-VZV gE IgG antibody concentration for which the response rate in the VV group is 95% or higher.
Percentage of participants reporting each solicited administration site event | Day 1 (post-dose) to Day 4
  Solicited administration site events include injection site redness, pain and swelling.
Percentage of participants reporting each solicited systemic event | Day 1 (post-dose) to Day 15
  Solicited systemic events include drowsiness, loss of appetite and irritability.
Percentage of participants reporting each solicited systemic event in terms of fever | Day 1 (post-dose) to Day 22
  Fever is defined as temperature greater than or equal to (>=)38.0 degrees Celsius (°C) by any route (the preferred location for measuring temperature is the axilla).
Percentage of participants reporting each solicited administration site event | Day 1 (post-dose) to Day 43
  Solicited administration site events include injection site varicella-like rash.
Percentage of participants reporting each solicited systemic event | Day 1 (post-dose) to Day 43
  Solicited systemic events include varicella-like rash (non-injection site) and general rash (not varicella-like).
Percentage of participants reporting unsolicited adverse events (AEs) | Day 1 (post-dose) to Day 43
  Unsolicited AEs include any AE reported in addition to solicited events during the study, or any "solicited" symptoms with onset outside of the specified period of follow-up for solicited symptoms, are assessed for each group after the administration of all vaccines.
Percentage of participants reporting medically attended AEs (MAAE) | Day 1 (post-dose) to Day 181 (study end)
  A MAAE is an AE for which the participant received medical attention including any symptom or illness requiring hospitalization, or an emergency room visit, or visit to/by a healthcare professional.
Percentage of participants reporting serious adverse events (SAEs) | Day 1 (post-dose) to Day 181 (study end)
  A SAE is an AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or other situations that are considered serious per medical or scientific judgment.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, Layton, Utah

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf